CLINICAL TRIAL: NCT00147992
Title: Immediate Loading of Implants in Totally Edentate Upper and Lower Jaw. A Retrospective Trial to Evaluate Survival of the Implants and Bridges, Quality of Prosthetic Work and Patient Satisfaction
Brief Title: Immediate Loading of Implants in Totally Edentate Upper and Lower Jaw. Trial to Evaluate Survival of the Implants and Bridges, Quality of Prosthetic Work and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/133
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2015-06

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- implants (Experimental)
  Interventions: Procedure: Immediate loading of implants in totally edentate upper and lower jaw

INTERVENTIONS:
Procedure: Immediate loading of implants in totally edentate upper and lower jaw — Immediate loading of implants in totally edentate upper and lower jaw.

SUMMARY:
This study is an evaluation of the survival of the implants and bridges, quality of prosthetic work and patient satisfaction after immediate loading of the implants in a totally edentate upper and lower jaw.

DETAILED DESCRIPTION:
This study is an evaluation of the survival of the implants and bridges, quality of prosthetic work and patient satisfaction after immediate loading of the implants in a totally edentate upper and lower jaw.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old

Exclusion Criteria:

* Medical risk patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Survival of implants and bridges | At beginning until last follow up

SECONDARY OUTCOMES:
Quality of prosthetic work | At end of follow up
Patient satisfaction | At end of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be